CLINICAL TRIAL: NCT04234451
Title: Efficacy, Safety and Underlying Mechanisms of Sphenopalatine Ganglion Acupuncture for Perennial Allergic Rhinitis: a Randomized, Double-blind, Placebo Controlled Study
Brief Title: Efficacy, Safety and Underlying Mechanisms of Sphenopalatine Ganglion Acupuncture for Perennial Allergic Rhinitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPA acupuncture for PAR
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Perennial Allergic Rhinitis
Keywords: Acupuncture; sphenopalatine ganglion; perennial allergic rhinitis; neuropeptides; inflammatory cytokines; neuro-immune interactions
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPA acupuncture (Active Comparator): active SPG acupuncture plus rescue medication (AA group)
  Interventions: Procedure: SPA acupuncture
- sham acupuncture (Sham Comparator): sham-SPG acupuncture plus rescue medication (SA group)
  Interventions: Procedure: sham acupuncture

INTERVENTIONS:
Procedure: SPA acupuncture — For patients in the AA group, acupuncture was performed at a selected point in the SPG by inserting the needle from the lower border of the zygomatic arch, posterior to the suture protuberance between the zygomatic process and temporal process. The needle was directed obliquely anteriorly, until nearly the whole needle was beneath the skin, and then rotated until the patient felt "de-qi" sensations . The patients in the AA group received four courses of active acupuncture(visit 1,2,3 and 4), twice a week during weeks 1 and 2, and then followed-up for a further 2 weeks (visit 5 during week 3 and visit 6 during week 4).
  Arms: SPA acupuncture
Procedure: sham acupuncture — For patients in the SA group, the needle was inserted at the same acupuncture point as for patients in the AA group, but to a depth of only 2-3cm and the procedure of rotating, twirling and thrusting the needle was repeated. During the acupuncture process, the acupuncturist sat on the side of the participant, where the patient could neither see the acupuncturist's face nor the length of the needle. The patients in the SA group received four courses of active acupuncture(visit 1,2,3 and 4), twice a week during weeks 1 and 2, and then followed-up for a further 2 weeks (visit 5 during week 3 and visit 6 during week 4).
  Arms: sham acupuncture

SUMMARY:
In recent years, a number of randomized controlled trials have confirmed the efficacy and safety of acupuncture in the treatment of allergic rhinitis (AR). Indeed, the latest American clinical guidelines recommended acupuncture treatment for AR patients who are interested in non-pharmacological treatment.

In conventional acupuncture treatment for AR, needles are inserted at specific acupoints in the body; with several studies demonstrating acupuncture of sphenopalatine ganglion (SPG) to improve nasal symptoms and quality of life in nasal inflammatory diseases.

The investigators hypothesize that, compared with sham acupuncture and rescue medication (RM), active SPG acupuncture combined with RM would lead to greater improvements in symptoms score and reduction in overall need for antihistamines. To test this hypothesis the investigators design a randomized, double blind, controlled trial to evaluate the efficacy of SPG acupuncture in perennial AR patients (allergic to indoor allergens, including house dust mite, fungi, animal dander and so one) and to explore the potential underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* 1. history of physician-diagnosed PAR with at least 2 years of typical symptoms
* 2. course on each onset lasting at least 4 weeks
* 3. skin prick test and/or serum antigen specific IgE positive to indoor allergens(sIgE≥0.7kU/L,≥class 2)
* 4. good patient compliance on acupuncture treatment
* 5. total nasal symptom scores(TNSS)>6 at V0

Exclusion Criteria:

* 1. oral steroids within 4 weeks prior to recruitment
* 2. nasal steroids and/or antihistamine 2 weeks prior to recruitment
* 3. seasonal AR
* 4. any respiratory infection within the previous 4 weeks prior to recruitment
* 5. history of nasal polyps, nasal septum deviation, asthma or autoimmune disorders
* 6. previously received acupuncture therapy for AR within 1 month prior to recruitment
* 7. women during pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline symptom scores at visit 4 | Symptom scores will be assessed at baseline (V0), visit 4( V4). V4 is at the second week 15 minutes after the fourth acupuncture.
  Patients recorded nasal and ocular symptom severity during the trial. Four nasal symptoms (itching, sneezing, rhinorrhoea and nasal obstruction) and two ocular symptoms (ocular itch and watery eyes) were individually graded on a ten-point scale (0, no symptoms; 1-3, mild symptoms; 4-7, moderate symptoms; 8-10, severe symptoms). Our primary outcome is total nasal symptom scores at Visit 4 (15 minutes after the fourth acupuncture ). The investigator will compare the symptom scores between the active acupuncture group and the sham acupuncture group.

SECONDARY OUTCOMES:
Rescue medication score | RMS will be assessed at baseline (V0), and each visit. V1, V2, V3, and V4 is on Day 1, Day 4, Day 8 and Day 11, respectively(+/- 1 day). V5 is at the third week and V6 is at the fourth week. There is no acupuncture during both V5 and V6.
  when the symptoms were very severe and could not be tolerated, the patients could use loratadine as rescue medication. The need for rescue medication was assessed as rescue medication score (RMS), analyzed as the weekly sum of daily use of Loratadine (10mg/d, equivalent to 1 point) or nasal corticosteroid spray (2 points)
rhinoconjunctivitis quality of life questionnaire (RQLQ) | RQLQ will be assessed at baseline (V0), and each visit. V1, V2, V3, and V4 is on Day 1, Day 4, Day 8 and Day 11, respectively(+/- 1 day). V5 is at the third week and V6 is at the fourth week. There is no acupuncture during both V5 and V6.
  RQLQ is assessed to evaluate the quality of life influenced by PAR. It offers 28 items related quality of life and each item ranges from 0 to 6, with lower scores implying a better health-related quality of life.
nasal patency | NCV, NAR and MCA will be assessed at baseline (V0), and each visit. V1, V2, V3, and V4 is on Day 1, Day 4, Day 8 and Day 11, respectively(+/- 1 day). V5 is at the third week, and V6 at the fourth week.
  Eccovision acoustic rhinometry (Hood Labs, Pembroke, USA) was used to measure the total nasal cavity volume (NCV) and minimum cross-sectional area (MCA). The ATMO 300 Rhinomanometer (ATMOS MedizinTechnikGmbH&Co., Feldkirch, Germany) was used to measure the nasal airway resistance (NAR) by anterior active rhinomanometry.
neuropeptides in nasal secretions | Nasal secretions can be obtained at baseline (V0), V4,V5 and V6. V4 is at the second week. V5 is at the third week and V6 is at the fourth week. There is no acupuncture during both V5 and V6.
  The levels of neuropeptides; including substance P, vasoactive intestinal peptide (VIP) , neuropeptide Y (NPY)) will be analysed using ELISA. The unit of all these parameters is ng/ml.
inflammatory cytokines in nasal secretions | Nasal secretions can be obtained at baseline (V0), V4 ,V5 and V6. V4 is at the second week. V5 is at the third week and V6 is at the fourth week. There is no acupuncture during both V5 and V6.
  The levels of inflammatory cytokines; including interferon-γ (IFN-γ), tumor necrosis factor-α(TNF-α), interleukin (IL)-5, IL-8, IL-17A, and eotaxin in the supernatants will be analyzed using the Luminex System. The unit of all these parameters is pg/ml.
adverse events | adverse events will be recorded at baseline (V0), and each visit. V1, V2, V3, and V4 is on Day 1, Day 4, Day 8 and Day 11, respectively(+/- 1 day). V5 is at the third week and V6 is at the fourth week. There is no acupuncture during both V5 and V6.
  Any adverse event following acupuncture was assessed by physicians and patients. Patients were instructed to record any unexpected signs, symptoms, and feelings during the entire trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi SM, Park JE, Li SS, Jung H, Zi M, Kim TH, Jung S, Kim A, Shin M, Sul JU, Hong Z, Jiping Z, Lee S, Liyun H, Kang K, Baoyan L. A multicenter, randomized, controlled trial testing the effects of acupuncture on allergic rhinitis. Allergy. 2013 Mar;68(3):365-74. doi: 10.1111/all.12053. Epub 2012 Dec 18. PMID 23253122
- [Background] Xue CC, Zhang AL, Zhang CS, DaCosta C, Story DF, Thien FC. Acupuncture for seasonal allergic rhinitis: a randomized controlled trial. Ann Allergy Asthma Immunol. 2015 Oct;115(4):317-324.e1. doi: 10.1016/j.anai.2015.05.017. Epub 2015 Jun 11. PMID 26073163
- [Background] Wang K, Chen L, Wang Y, Wang C, Zhang L. Sphenopalatine Ganglion Acupuncture Improves Nasal Ventilation and Modulates Autonomic Nervous Activity in Healthy Volunteers: A Randomized Controlled Study. Sci Rep. 2016 Jul 18;6:29947. doi: 10.1038/srep29947. PMID 27425415
- [Background] Brinkhaus B, Ortiz M, Witt CM, Roll S, Linde K, Pfab F, Niggemann B, Hummelsberger J, Treszl A, Ring J, Zuberbier T, Wegscheider K, Willich SN. Acupuncture in patients with seasonal allergic rhinitis: a randomized trial. Ann Intern Med. 2013 Feb 19;158(4):225-34. doi: 10.7326/0003-4819-158-4-201302190-00002. PMID 23420231